CLINICAL TRIAL: NCT03362489
Title: Conversion of in Vitro Fertilization Cycles to Intrauterine Inseminations in Patients With a Poor Ovarian Response to Stimulation
Acronym: ConFIRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-A00862-51
Record Dates: First submitted 2017-11-24; First posted 2017-12-05 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Infertility
Keywords: In Vitro Fertilization; Intra-Uterine Insemination; Poor responders
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVF / IVF-ICSI (Other): In Vitro Fertilization / In Vitro Fertilization - Intracytoplasmic Sperm Injection (ICSI)
  Interventions: Procedure: IVF / IVF-ICSI
- IUI (Other): Intrauterine insemination
  Interventions: Procedure: IUI

INTERVENTIONS:
Procedure: IVF / IVF-ICSI — In the "IVF" arm, oocyte retrieval is performed 36 hours after the HCG injection, in the operating room, under transvaginal ultrasound guidance, under local or general anesthesia. The procedure lasts about 20 minutes and the patients are discharged on the same day. The oocytes retrieved from the follicles are transported immediately to the lab for fertilization with the partner's sperm. Fertilization is done either via conventional IVF, or via ICSI, depending on the indication. Embryos are later transferred into the uterus on day 3 or day 5, under ultrasound guidance, in the outpatient department.
  Arms: IVF / IVF-ICSI
Procedure: IUI — In the "conversion to IUI" arm, IUI is performed 24 to 36 hours after ovulation trigger. The partner provides the sperm on site on the morning of the insemination, which is performed in the outpatient department.
  Arms: IUI

SUMMARY:
The purpose of this study is to compare the efficiency of conversion to IUI and IVF in patients with a poor ovarian response to stimulation

DETAILED DESCRIPTION:
In 5 to 10% of in vitro fertilization (IVF) cycles, a poor response to ovarian stimulation (defined as less than 4 mature follicles) is noted, even though high doses of exogenous gonadotropins are used. To date, there is no consensus on the ideal management strategy in poor responders. There are three therapeutic options available nowadays:

1. Oocyte retrieval is performed and the IVF cycle continued, despite the low number of mature follicles.
2. Conversion of the IVF cycle to an intrauterine insemination (IUI), on the condition of having at least one patent fallopian tube and good semen parameters.
3. Cancelation of the IVF cycle. In everyday practice, it is difficult for the physician to cancel the IVF cycle in the presence of 2, 3 or 4 mature follicles, especially following a lengthy stimulation.

If live birth rates were comparable between IUI and IVF, conversion to IUI would be the better option for poor responders, since it would avoid an invasive procedure (oocyte retrieval) and the associated risk of complications, and is associated with at a lower cost.

To our knowledge, no prospective randomized controlled trial comparing IVF to conversion to IUI in poor responders has been published to date. The studies published so far have been retrospective and observational, and had several methodological flaws.

Therefore, we aimed to analyze whether conversion of IVF cycles to IUI in poor responders would result in the same live birth rates as oocyte retrievals followed by embryo transfers.

ELIGIBILITY:
Inclusion Criteria:

* Patients who accepted being included and signed the consent forms.
* Age ≥18 years et <43 years.
* IVF cycle with and without Intra Cytoplasmic Sperm Injection (ICSI):

  * "Conventional" Agonist (long and short) or antagonist protocol, using urinary or recombinant gonadotropins.
  * Having only 2, 3 or 4 mature follicles (≥14 mm) on ovulation trigger day.

Exclusion Criteria:

* Confirmed bilateral tubal occlusion
* Non-French speaking patients
* Partners with severe oligoasthenoteratospermia (OATS) (<5 millions motile spermatozoa in the ejaculate)
* Suboptimal stimulation protocols:

  * Protocols ≤ 150 IU of daily gonadotropins
  * Mild stimulation protocols
  * Natural and modified natural cycle protocols
* Women under legal guardianship
* Women with no health or social security coverage
* Women participating in other interventional trials

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 462 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
The main criterion is the live birth rate | 12 months
  Defined as the birth of a living infant after 22 weeks gestational age (GA), or weighing ≥ 500 g.

SECONDARY OUTCOMES:
Biochemical pregnancy rate | 5 Weeks
  Defined as serum HCG levels >10 IU/L, 14 days after the IUI or the embryo transfer, followed by a rapid decrease until being undetectable.
Clinical pregnancy rate | 6-7 Weeks
  Defined as fetal cardiac activity at 6-7 weeks GA
Spontaneous pregnancy loss (PL) rate | 12 Weeks
  Including early and late pregnancy losses
Multiple pregnancy rate | 7-8 Weeks
  Defined as more than two embryos visualized on ultrasound at 7 weeks GA.
Term at delivery | 12 Months
  Term at delivery in Gestational age (GA)
Neonatal complications | 12 Months
  Neonatal complications
Neonatal survival | 12 Months
  Neonatal survival
All outcome measure will be further analyzed according to the number of follicles on trigger day (2, 3 or 4) and patients' age (<40 years vs. ≥40 years) | 12 Months
  Assess the impact of conversion to IUI, compared to IVF, on overall outcomes in in women with a poor ovarian response to stimulation, according to the number of follicles on trigger day (2, 3 or 4) and patients' age (<40 years vs. ≥40 years)
All outcome measures will be further analyzed in the subgroup of women considered poor responders according to the Bologna criteria | 12 Months
  Assess the clinical efficiency of conversion to IUI, compared to IVF, in women considered "poor ovarian responders" according to the Bologna criteria
The rate of IVF cycles with empty follicle syndrome and no embryo transfers. | 1 Week
  Analyze the rate of IVF cycles with empty follicle syndrome and no embryo transfers
Cumulative clinical pregnancy and live birth rates in the IVF group, thus taking into account fresh and frozen embryos transferred in subsequent cycles | 12 Months
  Assess the impact of conversion to IUI, compared to IVF, on the cumulative clinical pregnancy and live birth rates - taking into account frozen embryo transfers in IVF - in women with a poor ovarian response to stimulation
Cost-efficiency analysis at 12 months | 12 Months
  Compare the cost-efficiency of both strategies at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Emmanuel BOUET, MD, Study Director — University Hospital of Angers
Locations (32):
- France (31):
  - Victor Pauchet Clinic, Amiens
  - UH Angers, Angers
  - UH Besançon, Besançon
  - Jean Verdier Hospital, APHP, Bondy
  - Polyclinique Jean Villar, Bruges
  - UH Caen, Caen
  - Clinique Léonard de Vinci, Chambray-lès-Tours
  - Cholet Hospital, Cholet
  - Antoine Béclère Hospital AP-HP, Clamart
  - Sud Francilien Hospital, Corbeil-Essonnes
  - IHC Créteil, Créteil
  - UH Grenoble, Grenoble
  - Tertre Rouge Clinic, Le Mans
  - UH Lille, Lille
  - Lorient Hospital, Lorient
  - UH La conception AP-HM, Marseille
  - Clinique Jules Verne, Nantes
  - UH Nantes, Nantes
  - Clinique Pierre Cherest, Neuilly-sur-Seine
  - UH Nîmes, Nîmes
  - Hospital of Orléans, Orléans
  - Cochin Hospital, APHP, Paris
  - Poissy Saint Germain en Laye Hospital, Poissy
  - UH Potiers, Potiers
  - Clinique Mutualiste de la Sagesse, Rennes
  - UH Rennes, Rennes
  - UH Rouen, Rouen
  - Polyclinique de L'Atlantique, Saint-Herblain
  - UH Strasbourg, Strasbourg
  - UH Toulouse, Toulouse
  - UHR Tours, Tours
- UH Pointe-à-Pitre, Pointe-à-Pitre, Guadeloupe/France, Guadeloupe

REFERENCES:
- [Derived] Delbos L, Parot-Schinkel E, El Hachem H, Legendre G, Descamps P, Boucret L, Ferre-L'Hotellier V, Jeanneteau P, Dreux C, Moriniere C, May-Panloup P, Bouet PE. ConFIRM trial - conversion of in vitro fertilization cycles to intrauterine inseminations in patients with a poor ovarian response to stimulation: a protocol for a multicentric, prospective randomized trial. Trials. 2018 Oct 17;19(1):565. doi: 10.1186/s13063-018-2936-5. PMID 30333054